CLINICAL TRIAL: NCT00661063
Title: Diabetic Neuropathic Pain Topical Treatment- Comparative Study
Brief Title: Diabetic Neuropathy Topical Treatment
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Irmandade da Santa Casa de Misericordia de Sao Paulo (Other)
Responsible Party: Judymara Lauzi Gozzani PhD, ISCMSP
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 042/2007
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Last update posted 2008-04-18 (Estimated); Status verified 2008-04

CONDITIONS: Diabetic Neuropathy; Pain
Keywords: neuropathic pain; ketamine; clonidine; association
MeSH Terms: conditions — Diabetic Neuropathies; Pain; Neuralgia | interventions — Ketamine; Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- K (Experimental): drug - ketamine 1% gel
  Interventions: Drug: ketamine
- P (Placebo Comparator): vehicle gel
  Interventions: Drug: vehicle gel
- M (Experimental): association of ketamine and clonidine gel
  Interventions: Drug: ketamine + clonidine
- C (Experimental): clonidine gel
  Interventions: Drug: clonidine gel 1%

INTERVENTIONS:
Drug: ketamine — ketamine 150 mcg/g bid
  Arms: K
Drug: vehicle gel — bid - 12 weeks
  Arms: P
Drug: ketamine + clonidine — ketamine 150mcg/g + clonidine 1% gel bid 12 weeks
  Arms: M
Drug: clonidine gel 1% — bid 12 weeks
  Arms: C

SUMMARY:
Comparative study of efficacy and safety of ketamine, clonidine, mixture of both and placebo in patients with diabetic neuropathic pain

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus type I or II
* Mono or polyneuropathy
* Treatment with Tricyclic Antidepressant, Carbamazepine during 3 weeks at least
* Preserved cognition

Exclusion Criteria:

* Ulcerative or infection or vesicle lesion in pain site
* Pregnancy
* Breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-04 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
pain evaluation by visual analogue scale | 12 weeks

SECONDARY OUTCOMES:
pain evaluation by amount of rescue medication required | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Judymara L Gozzani, Investigator, Principal Investigator — Santa Casa de São Paulo
Locations (1):
- Santa Casa de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Serednicki WT, Wrzosek A, Woron J, Garlicki J, Dobrogowski J, Jakowicka-Wordliczek J, Wordliczek J, Zajaczkowska R. Topical clonidine for neuropathic pain in adults. Cochrane Database Syst Rev. 2022 May 19;5(5):CD010967. doi: 10.1002/14651858.CD010967.pub3. PMID 35587172